

## **PROTOCOL**

**Overview.** We conducted a pilot randomized controlled trial (RCT) that compared a prototype of MBTA to aa active control condition. We collected data at baseline and at follow-up (three-months later). Participants in the active control condition did not receive the MBTA prototype until the follow-up assessment. Aims of the study were to evaluate the feasibility, acceptability, and preliminary effectiveness of the MBTA prototype in promoting Veterans' support-seeking in a sample of recently separated Veterans. Findings will be used to guide further modifications to MBTA, as this pilot study used a prototype of MBTA.

Sampling and Data Collection Method. We drew participants from a sampling frame of recently separated Veterans identified from the VA/DoD Identity Repository (VADIR). VADIR maintains automated files on all former military personnel with the necessary demographic and military background information to support the study. Inclusion criteria was: (1) having separated from active duty military service within the past year but not the past three months (for whom not enough time may have gone by to adequately assess readjustment challenges); (2) having a postal address in the U.S; (3) having access to the internet; and (4) having an honorable discharge from the military. We sent 500 initial invitations to potential participants, with the goal of obtaining a sample of 106 Veterans at baseline. Twenty-five invitations were undeliverable. We applied a modification of the Dillman mail survey. Specifically, a VA-approved vendor mailed an invitation letter to potential participants, along with information about how to complete the study at a secure website. Veterans were randomly assigned to the intervention or active control condition prior to mailing. Consistent with Dillman's recommendation for repeated contacts, a reminder letter was mailed, followed by a second reminder letter, and then a final reminder letter at the first (T1; baseline) and second (T2; three-month follow-up) wave of data collection. We sent a final mailing with a monetary incentive in the form of a \$25 Amazon gift card to Veterans who completed T1 (baseline) and increased the incentive to \$50 at T2 (three-month follow-up). The informed consent process was administered electronically. Informed consent elements were displayed on the screen along with a button that potential participants could select to consent to participate. Participants had the option to print the page and/or request a copy from the research team. A total of 43 Veterans elected to participate in this study and provided data at baseline.

Intervention Approach. This MBTA prototype required Veterans to complete a 6-8 minute online assessment that measured areas of unmet well-being and mental health needs, after which they received individualized feedback on areas of unmet need, along with tailored recommendations for relevant programs, services, and supports. Veterans assigned to the intervention condition completed MBTA at T1 (baseline); Veterans in the active control condition had the opportunity to complete MBTA at T2 (three-month follow-up). Drawing on recommendations from the feedback-informed treatment (FIT) literature, MBTA feedback was provided via a brief, easy-to-read infographic that included recommendations for relevant resources. The research team generated a list of vetted resources that were free to use and nationally available prior to study. Relevant context was provided to normalize readjustment challenges and feedback was framed in terms of response formats rather than peer comparisons. For example, within the domain of financial satisfaction Veterans received the feedback that they indicated not being satisfied with their finances on average, rather than that they are less satisfied than their peers. Because the report was provided online it was possible to present information in an easily digestible manner, for example, by limiting the amount of information presented on each page and providing feedback in tabs rather than a list-based format. We also offered Veterans the opportunity to download a printable version of the report for future use.

## STATISTICAL ANALYSIS PLAN

For primary outcome #1, we generated frequency statistics. Primary analyses #2 and #3 involved evaluating the feasibility and acceptability of the tool (i.e., primary outcomes labeled as satisfaction of the tool) through qualitative data analysis of open-ended questions, specifically rapid content analysis. Unfortunately, the clincialtrials.gov platform does not allow reporting on these types of analyses. Thus, the primary analyses that are presented here reflect only a subset of the analyses that were the focus of this study. We provided counts of themes generated from our qualitative data analysis.

For our secondary outcomes, specifically #1, #3, and #4, ANCOVA models were run. Baseline scores of the construct of interest and group status (intervention or active control) were entered as the independent variables and follow-up scores of the construct of interest was entered as the dependent variable. We also found significant age differences between the intervention and active control group, and differences among constructs of interest at baseline by age, so age was also entered in the models as a covariate. Due to the small sample size of this pilot study, we encourage readers to focus on the magnitude of the effect that are provided in the results, specifically partial eta-squared values:  $\eta 2 = 0.01$  indicate a small effect;  $\eta 2 = 0.06$  indicate a medium effect;  $\eta 2 = 0.14$  indicate a large effect. This study was not powered to detect statistically significant differences, although this information is presented due to clinicaltrial gov requirements.

For our secondary outcome #2, frequency statistics are reported. Participants who did not report challenges within a domain could not be categorized into a stage of change; therefore, our sample size for these analyses are smaller than the other secondary outcomes. Due to the smaller than expected sample size and because chi-square tests are sensitive to sample size, we elected to report descriptive information only for this outcome. We examined the subset of participants that reported challenges within a domain at baseline and then examined if they moved forward in their stages of change/were taking action to address these challenges by the three month-follow-up.

**For our secondary outcome #5, we generated frequency statistics.** Specifically, the number of participants that reported the MBTA prototype increased their awareness, encouraged them to improve their well-being, and if the Veteran reported using a resource/service. For the specific types of services used, frequency statistics were limited to the subset of Veterans that reported using a resource/service between baseline and follow-up.